CLINICAL TRIAL: NCT02783690
Title: A Randomized Trial of 15 Fraction vs 25 Fraction Pencil Beam Scanning Proton Radiotherapy After Mastectomy in Patients Requiring Regional Nodal Irradiation
Brief Title: A Trial of 15 Fraction vs 25 Fraction Pencil Beam Scanning Proton Radiotherapy After Mastectomy in Patients Requiring Regional Nodal Irradiation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-006137; MC1631 (Other: Mayo Clinic); NCI-2017-02362 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCT03391453 (obsolete NCT alias)
Record Dates: First submitted 2016-05-19; First posted 2016-05-26 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Fractionation (No Intervention): 50.0 Gy (RBE) in 25 daily fractions
- Hypofractionation (Experimental): 40 Gy (RBE) in 15 daily fractions
  Interventions: Radiation: Hypofractionation

INTERVENTIONS:
Radiation: Hypofractionation — 40 Gy (RBE) in 15 daily fractions
  Arms: Hypofractionation

SUMMARY:
This is a randomized controlled trial to determine the safety of 15 fraction vs 25 fraction pencil beam scanning proton radiotherapy after mastectomy in patients requiring regional nodal irradiation. Proton therapy is recognized as a standard option for the delivery of radiotherapy for breast cancer.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years
* Histologic confirmation of breast cancer resected by mastectomy with or without immediate reconstruction and chest wall and regional nodal irradiation planned.
* pStage T1-T4N0-N3M0 or ypStage T0-4N0-N3M0 Note: The axilla must be staged by sentinel node biopsy alone, sentinel node biopsy followed by axillary node dissection, or axillary lymph node dissection alone
* ECOG Performance Status (PS) 0 to 2. (Appendix I).
* Negative pregnancy test done ≤7 days prior to registration, for women of childbearing potential only.
* Radiotherapy must begin within 12 weeks of last surgery (breast or axilla) or last chemotherapy.

Note: Breast implants and expanders allowed

* Able to and provides IRB approved study specific written informed consent
* Ability to complete questionnaire (s) by themselves or with assistance
* Able to complete all mandatory tests listed in section 4.0
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide tissue and blood samples for correlative research purposes.
* Rochester and Arizona patients: Willing to sign consent onto the Mayo Clinic Radiotherapy Patient Outcomes Registry and Biobanking study, IRB number 15-000136
* Rochester patients: Willing to sign consent onto Evaluation of cardiac function in patients undergoing proton beam or photon radiotherapy, IRB number 15-007443

Exclusion Criteria:

* Medical contraindication to receipt of radiotherapy.
* Severe active co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or providing informed consent.
* Active systemic lupus or scleroderma.
* Pregnancy or women of childbearing potential who are sexually active and not willing/able to use medically acceptable forms of contraception
* Prior receipt of ipsilateral breast or chest wall radiation that would result in significant overlap of radiation therapy fields. Prior contralateral radiotherapy for breast cancer is allowed.
* Positive margins after definitive surgery
* History of non-breast malignancies (except for in situ cancers treated only by local excision and basal cell and squamous cell carcinomas of the skin) within 5 years prior study entry
* Inflammatory breast cancer
* Recurrent Breast Cancer
* Boosts to the chest wall after mastectomy. Nodal boosts are allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2023-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W. Mutter, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- [Derived] Mutter RW, Giri S, Fruth BF, Remmes NB, Boughey JC, Harless CA, Ruddy KJ, McGee LA, Afzal A, Gao RW, Shumway DA, Vern-Gross TZ, Villarraga HR, Kenison SL, Kang Y, Wong WW, Stish BJ, Merrell KW, Yan ES, Park SS, Corbin KS, Vargas CE. Conventional versus hypofractionated postmastectomy proton radiotherapy in the USA (MC1631): a randomised phase 2 trial. Lancet Oncol. 2023 Oct;24(10):1083-1093. doi: 10.1016/S1470-2045(23)00388-1. Epub 2023 Sep 8. PMID 37696281
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypofractionation: 40 Gy (RBE) in 15 daily fractions> Hypofractionation: 40 Gy (RBE) in 15 daily fractions
Period: Overall Study
Arm/Group | Conventional Fractionation | Hypofractionation
Started | 44 | 44
Completed | 41 | 41
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Fractionation | Hypofractionation | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Continuous [Median (Full Range); unit: years] | 50 [30 to 76] | 54 [32 to 78] | 52 [30 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 82
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 38 | 41 | 79
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 40 | 39 | 79
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Complication Rate
Description: Will be defined as the percentage of women randomized who develop one or more of the following events: grade 3 or higher late adverse events; unplanned surgical intervention (not including planned serial fat grafting) in patients who undergo mastectomy with reconstruction.
Time Frame: 24 months
Population: All treated patients were included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Fractionation | Hypofractionation
Number analyzed (Participants) | 41 | 41
percentage of participants | 15 | 20

2. Secondary Outcome: Incidence of Acute Adverse Events
Description: Acute adverse events are defined using Common Terminology Criteria for Adverse Events (CTCAE) version 4. Grade 1 or 2 events occurring in at least 10% of patients are reported along with all grade 3 or higher events.
Time Frame: 5 years
Measure: Number; unit: event occurrence
Arm/Group | Conventional Fractionation | Hypofractionation
Number analyzed (Participants) | 41 | 41
event occurrence
  Breast infection | 1 | 3
  Oesophagitis | 5 | 8
  Breast oedema | 9 | 4
  Skin hyperpigmentation | 32 | 21
  Oedema of the limbs | 5 | 2
  Radiation dermatitis | 39 | 40
  Stroke | 0 | 1
  Non-cardiac chest pain | 2 | 2
  Joint range of motion decreased | 11 | 7

3. Secondary Outcome: Incidence of Late Adverse Events
Description: Late adverse events are defined using CTCAE version 4. Grade 1 or 2 events occurring in at least 10% of patients are reported along with all grade 3 or higher events.
Time Frame: 5 years
Population: All patients that were evaluated for adverse events 90 or more days after radiotherapy.
Measure: Number; unit: event occurrence
Arm/Group | Conventional Fractionation | Hypofractionation
Number analyzed (Participants) | 40 | 40
event occurrence
  Breast infection | 0 | 5
  Breast oedema | 3 | 10
  Skin hyperpigmentation | 19 | 22
  Joint range of motion decreased | 11 | 12
  Oedema of the limbs | 6 | 10
  Radiation dermatitis | 3 | 6
  Non-cardiac chest pain | 6 | 11
  Superficial soft tissue fibrosis | 5 | 7
  Fibrosis deep connective tissue | 10 | 7

4. Secondary Outcome: Reconstruction Failure
Description: A failure is defined as loss of the tissue expander or implant with the inability to replace it resulting in no final reconstruction or conversion to autologous reconstruction or revised with the addition of autologous reconstruction.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Fractionation | Hypofractionation
Number analyzed (Participants) | 41 | 41
Participants | 1 | 5

5. Secondary Outcome: Quality of Life - Breast Cancer Outcomes
Description: measured by cosmesis evaluation and the Breast Cancer Treatment Outcome Scale (BCTOS)
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2026-01

6. Secondary Outcome: Cosmesis
Description: measured by reviewing digital photographs and the 4 point (excellent, good, fair, poor) adaptation of the Harvard Cosmesis Scale
Time Frame: baseline, 2 years, and 5 years
Reporting Status: Not Posted

7. Secondary Outcome: Ipsilateral Breast Tumor Recurrence (IBTR) Incidence
Description: Will be defined as local recurrence from trial registration as a first event at 5 years. The IBTR cumulative incidence will be estimated using a competing risks method by treatment arm. The competing risks will be regional/distant breast cancer recurrence and death. The percentage of patients with IBTR is defined as the number of patients that have a IBTR divided by the number of patients treated in each arm.
Time Frame: 5 years
Measure: Number; unit: percentage of patients
Arm/Group | Conventional Fractionation | Hypofractionation
Number analyzed (Participants) | 41 | 41
percentage of patients | 0 | 2

8. Secondary Outcome: Distant Recurrence Incidence
Description: Will assess metastatic cancer that has either been biopsy confirmed or clinically diagnosed as recurrent invasive breast cancer at 5 years. The percentage of patients with a distant recurrence is defined as the number of patients that have a distant recurrence divided by the number of patients treated in each arm.
Time Frame: 5 years
Measure: Number; unit: percentage of patients
Arm/Group | Conventional Fractionation | Hypofractionation
Number analyzed (Participants) | 41 | 41
percentage of patients | 10 | 7

9. Secondary Outcome: Regional Recurrence Incidence
Description: Defined as invasive breast cancer in the axilla, regional lymph nodes, chest wall, and skin of the ipsilateral breast at 5 years. The percentage of patients with a regional recurrence is defined as the number of patients that have a regional recurrence divided by the number of patients treated in each arm.
Time Frame: 5 years
Measure: Number; unit: percentage of patients
Arm/Group | Conventional Fractionation | Hypofractionation
Number analyzed (Participants) | 41 | 41
percentage of patients | 0 | 2

10. Secondary Outcome: Disease-free Survival (DFS) at 3 Years
Description: DFS is defined as the time from study registration until the occurrence, if any, of one of the following events: invasive IBTR, regional invasive breast cancer recurrence, distant breast cancer recurrence, death due to any cause, contralateral invasive breast cancer, and second primary non-breast invasive disease. DFS at 3 years will be reported as the percent of patients without a DFS event at 3 years post radiotherapy.
Time Frame: 3 years post radiotherapy, up to 38 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Conventional Fractionation | Hypofractionation
Number analyzed (Participants) | 41 | 41
percentage of patients | 89.4 [80.0 to 99.8] | 92.4 [84.5 to 100]

11. Secondary Outcome: Overall Survival (OS) at 3 Years
Description: Overall survival is defined as the time from registration to death due to any cause. OS at 3 years is reported as the percentage of patients still alive and in follow up at 3 years post radiotherapy.
Time Frame: 3 years post radiotherapy, up to 38 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Conventional Fractionation | Hypofractionation
Number analyzed (Participants) | 41 | 41
percentage of patients | 94.9 [88.2 to 100] | 95.1 [88.6 to 100]

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Conventional Fractionation | Hypofractionation
All-Cause Mortality (participants affected / at risk) | 2/44 | 2/44
Serious Adverse Events (participants affected / at risk) | 2/44 | 3/44
Other Adverse Events (participants affected / at risk) | 41/44 | 41/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Fractionation (N=44) | Hypofractionation (N=44)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Fractionation (N=44) | Hypofractionation (N=44)
Telangiestasia (Nervous system disorders) | 10 (285) | 8 (135)
Esophagitis (Gastrointestinal disorders) | 5 (6) | 8 (9)
Edema limbs (General disorders) | 10 (13) | 10 (17)
Non-cardiac chest pain (General disorders) | 8 (10) | 13 (17)
Breast infection (Infections and infestations) | 3 (3) | 7 (7)
Dermatitis radiation (Injury, poisoning and procedural complications) | 39 (45) | 40 (52)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 10 (14) | 7 (9)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 15 (33) | 15 (25)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 5 (6) | 7 (8)
Brachial plexopathy (Nervous system disorders) | 0 (0) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 33 (68) | 29 (61)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Lymphedema (Vascular disorders) | 11 (16) | 12 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT02783690/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT02783690/ICF_001.pdf